CLINICAL TRIAL: NCT07380165
Title: Expanded Access Program (EAP) of Levacetylleucine for Ataxia-Telangiectasia (A-T)
Status: Temporarily not available | Type: Expanded Access
Sponsor: IntraBio Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: IB1001-EA3
Record Dates: First submitted 2026-01-23; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Ataxia-Telangiectasia (A-T)
Keywords: Ataxia-Telangiectasia; Louis Bar Syndrome
MeSH Terms: conditions — Ataxia Telangiectasia | interventions — acetylleucine

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Levacetylleucine — 1 gram levacetylleucine as granules in unit-dose packet. Investigational drug is administered as oral suspension, up to three times per day, based on body weight.
  Other Names: AQNEURSA; N-Acetyl-L-leucine

SUMMARY:
This expanded access program provides investigational levacetylleucine to patients with Ataxia-Telangiectasia who are not eligible for clinical trials and have no satisfactory alternative therapies.

DETAILED DESCRIPTION:
This expanded access program provides access to investigational drug, levacetylleucine, for eligible patients with Ataxia-Telangiectasia that are not eligible for other clinical trials, and a medical doctor has decided there is potential benefit outweighing the risk of receiving an investigational therapy based on the patient's medical history and program eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a genetically confirmed diagnosis of Ataxia-Telangiectasia, a rare and serious disease with no alternative approved treatments.
2. Patient and/or their legal representative signed a written informed consent and, if applicable, written assent.
3. Patient weighs ≥15 kg.
4. If female and of reproductive potential, the treating physician verified the patient is not pregnant prior to enrollment and will use adequate contraceptive methods to avoid pregnancy during and up to 7 days after participating in the program.
5. Patient resides in the United States at time of enrollment and throughout the duration of their participation in the EAP.

Exclusion Criteria:

1. Patient is enrolled in or early withdrew participation from a clinical trial with levacetylleucine for A-T.
2. Patient is pregnant, breastfeeding, or considering pregnancy.
3. Patient has a physical, cognitive, psychiatric condition, or an active or suspected malignancy that, in the judgment of the treating physician, may pose a safety risk or interfere with the patient's ability to comply with the EAP procedures.
4. Patient is receiving N-acetyl-DL-leucine or N-acetyl-D-leucine and is unwilling to stop use throughout the duration of their participation in the EAP.
5. Patient is receiving another investigational drug for any reason.

Sex: All
Age Groups: Child, Adult, Older Adult